CLINICAL TRIAL: NCT05314062
Title: Effect of Iron-enriched Aspergillus Oryzae Compared to Ferrous Sulfate on the Growth and Virulence of Common Enteric Pathogens
Brief Title: Effect of Iron Source on the Growth of Enteric Pathogens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Stephen R. Hennigar, Ph.D., Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 00002850
Record Dates: First submitted 2022-03-19; First posted 2022-04-06 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Iron Deficiency Anemia Treatment
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous sulfate (FeSO4) (Active Comparator): FeSO4 supplements containing 54 mg elemental iron
  Interventions: Dietary Supplement: FeSO4
- Ferrous sulfate-enriched Aspergillus oryzae (Ao iron) (Experimental): Ao iron supplements containing 54 mg elemental iron
  Interventions: Dietary Supplement: Ao iron

INTERVENTIONS:
Dietary Supplement: FeSO4 — 2 FeSO4 supplements containing 27 mg elemental iron/supplements (54 mg total iron)
  Arms: Ferrous sulfate (FeSO4)
Dietary Supplement: Ao iron — 2 Ao iron supplements containing 27 mg elemental iron/supplements (54 mg total iron)
  Arms: Ferrous sulfate-enriched Aspergillus oryzae (Ao iron)

SUMMARY:
The World Health Organization recommends daily iron supplementation for infants and children (6 months-12 years). Based on the low cost and high bioavailability and efficacy, ferrous sulfate is typically the first choice for supplementation and fortification. The recommended dose of iron is set high to deliver adequate absorbed iron due to low rates of dietary iron absorption, which is typically <10%. Thus, the majority of dietary iron is not absorbed and travels to the colon. Unabsorbed iron in the colon may select for enteric pathogens at the expense of beneficial commensal bacteria and increase infection risk, including the clinical incidence of diarrhea. The objective of this study is to compare the effects of iron as ferrous sulfate (FeSO4) or FeSO4-enriched Aspergillus oryzae (Ao iron) on the growth and virulence of common enteric pathogens using an in vitro fecal fermentation model. Stool samples will be collected from children following ingestion of an iron supplement as either FeSO4 or Ao iron. Stool samples will be spiked with common enteric pathogens and outcome measures will be determined following in vitro fecal fermentation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 5-12 y
* Willing to donate stool sample

Exclusion Criteria:

* Currently taking antibiotics
* Currently taking a vitamin and mineral supplement containing iron
* Wards of the state, including children in foster care

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Concentration of iron taken up by enteric pathogens | 0-24 hours
  Iron uptake of common enteric pathogens will be determined in stool following in vitro fecal fermentation.
Growth of enteric pathogens measured by optical density | 0-24 hours
  Growth of common enteric pathogens will be determined in stool following in vitro fecal fermentation.

SECONDARY OUTCOMES:
Gut microbiome composition and diversity | 0-24 hours
  Gut microbiome composition will be determined in stool following in vitro fecal fermentation using 16S rRNA gene sequencing.
Individual fecal short chain fatty acid (SCFA) concentration | 0-24 hours
  Individual SCFAs will be determined in stool following in vitro fecal fermentation by liquid chromatography-mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.